CLINICAL TRIAL: NCT03868371
Title: Acute Changes in the Mineral Metabolism After a High Phosphorous Containing Meal in Dialysis Patients - a Randomized Cross-over Trial
Brief Title: Acute Changes in the Mineral Metabolism After a High Phosphorous Containing Meal in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Ditte Hansen, Associate professor, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H-18063465
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Disease Stage 5; Mineral Metabolism Disorder
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. high - 2. low (Active Comparator): These are the patients receiving a high phosphorous containing meal in the first trial day, and a low phosphorous containing meal in the second trial day.
  Interventions: Dietary Supplement: High phosphorous containing meal; Dietary Supplement: Low phosphorous containing meal
- 1. low - 2. high (Active Comparator): These are the patients receiving a low phosphorous containing meal in the first trial day, and a high phosphorous containing meal in the second trial day.
  Interventions: Dietary Supplement: High phosphorous containing meal; Dietary Supplement: Low phosphorous containing meal

INTERVENTIONS:
Dietary Supplement: High phosphorous containing meal — A meal with a high phosphorous content
Dietary Supplement: Low phosphorous containing meal — A meal with a low phosphorous content

SUMMARY:
The purpose of the study is to investigate whether a high phosphorous containing meal causes acute changes in p-phosphate levels in patients with dialysis-dependent kidney failure.

DETAILED DESCRIPTION:
Disturbances in the mineral metabolism and especially the phosphate metabolism is associated with increased risk of cardiovascular disease and death in patients with kidney failure. In the healthy population the kidney compensates for a high phosphorous intake by increase renal excretion of phosphate, but this is not possible for patients with kidney failure. Due to this monitoring and controlling phosphate levels is an important clinical goal in treatment of kidney failure, and it is often achieved with a phosphorous poor diet and phosphate binders.

Currently this monitoring of the phosphate level is complicated by a poor understanding of how plasma phosphate acutely reacts to a phosphate rich meal. Often patients may have consumed a phosphate rich meal shortly before their blood test is taken, which may have an acute impact on the plasma phosphate level in the blood test and complicated the task of assessing their chronic phosphate levels.

To examine this problem, the investigators wish to conduct a randomized cross-over trial, where peritoneal dialysis patients are recruited and randomly assigned to consume either a meal either high or low in phosphate on the first day of trial and the opposite in the second.

With blood tests just before and during 5 hours after the meal, the investigators will examine plasma-phosphate levels as well as other blood parameters of importance to the mineral metabolism to determine, whether a meal rich in phosphate causes significant changes in these test parameters compared to a meal poor in phosphate.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Currently treated with peritoneal dialysis (APD or CAPD)
* Serum ionized calcium between 1.10 and 1.40 mmol/L for >3 months
* Plasma phosphate between 0.7 and 3.0 mmol/L for >3 months

Exclusion Criteria:

* Earlier parathyroidectomized
* Other conditions, which hinders the participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Difference in plasma phosphate in mmol/L at 5 specific times following a high-phosphate containing meal compared to a low-phosphate containing meal measured by analyzing of blood samples at each specific time. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.

SECONDARY OUTCOMES:
Changes in plasma phosphate in mmol/L in blood samples at 5 specific times following a high-phosphate meal or low-phosphate meal compared to levels of plasma phosphate at preceding specific times and differences in these changes. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Difference in serum ionized calcium at 5 specific times following a high-phosphate containing meal compared to a low-phosphate containing meal measured by analyzing of blood samples at each specific time. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Changes in serum ionized calcium in blood samples at 5 specific times following a high-phosphate meal or low-phosphate meal compared to levels of serum ionized calcium at preceding specific times and differences in these changes. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Difference in plasma PTH at 5 specific times following a high-phosphate containing meal compared to a low-phosphate containing meal measured by analyzing of blood samples at each specific time. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Changes in plasma PTH in blood samples at 5 specific times following a high-phosphate meal or low-phosphate meal compared to levels of plasma PTH at preceding specific times and differences in these changes. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Difference in plasma FGF-23 at 5 specific times following a high-phosphate containing meal compared to a low-phosphate containing meal measured by analyzing of blood samples at each specific time. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Changes in plasma FGF-23 in blood samples at 5 specific times following a high-phosphate meal or low-phosphate meal compared to levels of plasma FGF-23 at preceding specific times and differences in these changes. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Difference in plasma magnesium at 5 specific times following a high-phosphate containing meal compared to a low-phosphate containing meal measured by analyzing of blood samples at each specific time. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Changes in plasma magnesium in blood samples at 5 specific times following a high-phosphate meal or low-phosphate meal compared to levels of plasma magnesium at preceding specific times and differences in these changes. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Difference in plasma 1,25(OH)2 Vitamin D at 5 specific times following a high-phosphate containing meal compared to a low-phosphate containing meal measured by analyzing of blood samples at each specific time. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Changes in plasma 1,25(OH)2 Vitamin D in blood samples at 5 specific times following a high-phosphate meal or low-phosphate meal compared to levels of plasma 1,25(OH)2 Vitamin D at preceding specific times and differences in these changes. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Difference in T50 at 5 specific times following a high-phosphate containing meal compared to a low-phosphate containing meal measured by analyzing of blood samples at each specific time. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Changes in T50 in blood samples at 5 specific times following a high-phosphate meal or low-phosphate meal compared to levels of T50 at preceding specific times and differences in these changes. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.
Differences in levels between the groups of serum ionized calcium, plasma PTH, plasma FGF-23, plasma magnesium, plasma 1,25(OH)2 Vitamin D, T50 and plasma phosphate at specific times following either a high phosphate or low phosphate containing meal. | 5 hours
  The specific times are: Before consumption of the meal(time 0), and 1 hour, 2 hours, 3 hours and 5 hours after consumption of the meal.

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, PhD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark